CLINICAL TRIAL: NCT05000775
Title: The Influence of a Microbiome Immunity Formula on Alteration of Anthropometric and Glycemic Indices and Modulation of Gut Microbiome in Obese Young Individuals in Hong Kong: A Randomized, Double-blinded, Placebocontrolled Study.
Brief Title: The Influence of GNiib® in Obesity Management in Obese Young Individuals in Hong Kong.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Alice Pik Shan KONG, Professor, Medicine and Therapeutics, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20210615-001
Record Dates: First submitted 2021-08-02; First posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G-Niib (Experimental): G-NiiB®, a patent-protected microbiome immunity formula, composed of naturally occurring food-grade bacteria approved by health authorities, has been developed by a group of CUHK gastroenterology experts.
  Interventions: Dietary Supplement: G-Niib
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: G-Niib — G-NiiB®, a patent-protected microbiome immunity formula, composed of naturally occurring food-grade bacteria approved by health authorities, has been developed by a group of CUHK gastroenterology experts.
  Arms: G-Niib
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Obesity is a global epidemic, and is an important cardio-metabolic risk factor associated with many non-communicable diseases, such as coronary artery disease (CAD), diabetes and non-alcoholic fatty liver diseases (NAFLD) (1-6). In 2010, our team recruited a cohort of obese adolescents [mean age at baseline: 17.2 years, mean body mass index (BMI): 30.9 kg/m2] from school surveys (7). Our group has examined the impact of dietary intervention using low glycemic index (GI) diet to reduce body weight of adolescents. We have reported that participants in the low GI group had a significantly greater reduction in obesity indices namely waist circumference after 6 months of intervention compared to counterparts in usual diet counselling group. We recently conducted a phone interview of the participants and most, if not all, of them remained obese from self-reported body weight. Pharmacological treatment options for obese individuals are limited (8-10). Amassing evidence showed that the gut microbiota plays an important role in energy harvesting and lipid metabolism. Gut microbiota dysbiosis was repeatedly reported in patients with obesity (11-13). Studies in humanized mouse models suggest that the obese gut microbiota was more efficient in harvesting energy from diet and may be a causative factor in the pathogenesis of metabolic disorders, including obesity, type 2 diabetes and NAFLD (14). Therefore, modulation of microbiota might be a potential strategy for prevention and treatment of metabolic disorders. Microbial-based therapeutics such as probiotics, prebiotics, symbiotic or fecal microbiota transplantation have shown promising effect in improving host metabolic health (15, 16). Prebiotics consumption changes the composition of gut microbiota, alters levels of satietogenic gut peptides, decreases systemic inflammation, and improves insulin sensitivity and glucose tolerance (17). Supplementation of probiotics in overweight and obese individuals with probiotics reduces body weight and obesity indices (16, 18, 19). The use of probiotics also reduces intrahepatic triglyceride (IHTG) in patients with non-alcoholic steatohepatitis (20) and improves post-prandial glucose control in subjects with type 2 diabetes (21). G-NiiB®, a patent-protected microbiome immunity formula, composed of naturally occurring food-grade bacteria approved by health authorities, has been developed by a group of CUHK gastroenterology experts.

DETAILED DESCRIPTION:
Study Design:

This will be a 24-week randomized double-blinded placebo-controlled study on the effect of G-NiiB®, CU Medicine Immunity Microbiome Formula, on young obese individuals who exited from a randomized controlled interventional trial with dietary intervention with low GI diet for 12-month that was conducted in 2010 (NCT no. 01278563). This study protocol complies with the Declaration of Helsinki and ICH-GCP guideline.

Subjects and Methods:

Inclusion Criteria:

1. 281 obese adolescents who participated in the randomized controlled interventional trial with low GI index diet
2. Willingness to give written consent

Exclusion Criteria:

1. Subjects who are allergic to any ingredients listed in G-NiiB®, microbiome immunity formula.
2. Subjects with any condition that the investigator deems as a sound reason (e.g. active gastrointestinal diseases and malignancies) for disqualification from enrollment into the study.

Study Procedures:

At screening visit:

Anthropometric measurements, including body weight and height, waist and hip circumferences, percentage body fat by bioimpedance (23).

Questionnaires to document 1) demographic data including past medical and history, birth weight, 2) 3-day diet record using locally validated questionnaires (24) and 3) physical activity level/log sheet (IPAQ) ; 4) change of eating behavior and quality of life by eating disorders examinations (EDE) and 36-item short form survey (SF-36).

Pharmacist to record past and present medication history, including prescribed drugs, over-the-counter drugs and supplements, especially, 1) Subjects who have received antibiotics, antifungal, antiparasitic, or antiviral treatment within 12 weeks prior to study entry; 2) Subjects who plan to use antibiotic, antifungal, antiparasitic, or antiviral treatment during the study; 3) Subjects using proton pump inhibitor; 4) Present use of probiotics/nutritional supplements e.g., the use of replacement doses of Vitamin D, calcium supplements, and multi-vitamin tablet.

After an overnight fast of 8-10 hours, baseline blood tests will be sampled including plasma glucose, insulin, complete blood picture, renal and liver function tests, thyroid function test, lipid profiles, high sensitivity C-reactive protein (hs-CRP) (25). Additional 15ml of blood will be collected for PBMC isolation (22). Spot urine for albumin-creatinine ratio will be collected for detection of microalbuminuria (26). Various indexes of insulin resistance (HOMA-IR) and pancreatic beta-cell function (HOMA-beta) will be calculated from the homeostasis model assessment (27). Insulin secretion will be calculated from plasma glucose and insulin during various time points of OGTT.

Liver assessment by transient elastography (Fibroscan®), in which controlled attenuation parameter (CAP) will be used to detect liver steatosis while liver stiffness measurement (LSM) will be used to assess liver fibrosis (28).

Ultrasound scan for mesenteric fat, fatty liver and carotid intimal medial thickness will be performed (29, 30).

Stool for gut microbiota will be sampled. Blood for genetic studies (5ml), plasma (350 µL) and urine (500 µL) for metabolomics investigations will also be stored.

At randomization visit:

Participants will be randomly assigned to either intervention or control arms in 1:1 ratio. Allocation will be performed using block randomization with varying block sizes to maintain a good balance of subjects between the two arms and optimize allocation concealment throughout the subject recruitment period. A random sequence of grouping identifiers (I=intervention or C=control), based on computer-generated random codes will be prepared in advance by a statistician who is independent to arm allocation. The allocation sequence list will be password-protected and stored in a computer, and only be accessible to staff who is for arm allocation. The arm allocation of each participant will be assigned sequentially according to his/her sequence of enrolment and the corresponding group identifier in the prior prepared random sequence list. The research staff responsible for data collection will be blinded to the arm allocation.

All participants will be dispensed a 12-week supply of double-blinded study intervention or placebo products. Each participant will be given an administration log to record the daily intake of G-NiiB® or its placebo-control. Patient will be counselled to take one packet of the dispensed product once daily and record the time of ingestion and any adverse reactions in the logbook daily for a total of 24 weeks. Patient will be advised to take photo of the administration logbook within first week of enrollment into this study to ensure the log entry has been filled accurately. Patient will receive monthly phone calls from a pharmacist to ensure compliance of study product administration (31).

At interim study visit (at 12-week) All participants will be dispensed a 12-week supply of double-blinded study intervention or placebo products. Administration logbook will be checked by research staff. Adherence will be documented to compare the good adherence group and bad adherence group for the efficacy of the product provided. Good adherence is defined as missing not more than one daily dose of the product provided, while poor adherence is defined as missing two or daily dose of the product provided.

Anthropometric measurements, including body weight and height, waist and hip circumferences, percentage body fat by bioimpedance (23).

Questionnaires to document 1) demographic data including past medical and history, birth weight, 2) 3-day diet record using locally validated questionnaires (24) and 3) physical activity level/log sheet (IPAQ) ; 4) change of eating behavior and quality of life by eating disorders examinations (EDE) and 36-item short form survey (SF-36).

Pharmacist to record past and present medication history, including prescribed drugs, over-the-counter drugs and supplements, especially, 1) Subjects who have received antibiotics, antifungal, antiparasitic, or antiviral treatment within 12 weeks prior to study entry; 2) Subjects who plan to use antibiotic, antifungal, antiparasitic, or antiviral treatment during the study; 3) Subjects using proton pump inhibitor; 4) Present use of probiotics/nutritional supplements e.g., the use of replacement doses of Vitamin D, calcium supplements, and multi-vitamin tablet.

After an overnight fast of 8-10 hours, baseline blood tests will be sampled including plasma glucose, insulin, complete blood picture, renal and liver function tests, thyroid function test, lipid profiles, high sensitivity C-reactive protein (hs-CRP) (25). Additional 15ml of blood will be collected for PBMC isolation (22). Spot urine for albumin-creatinine ratio will be collected for detection of microalbuminuria (26). Various indexes of insulin resistance (HOMA-IR) and pancreatic beta-cell function (HOMA-beta) will be calculated from the homeostasis model assessment (27). Insulin secretion will be calculated from plasma glucose and insulin during various time points of OGTT.

Liver assessment by transient elastography (Fibroscan®), in which controlled attenuation parameter (CAP) will be used to detect liver steatosis while liver stiffness measurement (LSM) will be used to assess liver fibrosis (28).

Stool for gut microbiota will be sampled. Blood for genetic studies (5ml), plasma (350 µL) and urine (500 µL) for metabolomics investigations will also be stored.

At follow-up visit (at 24-week) Repeat study procedures at baseline visit. All the unused products must be returned to research team for examination.

ELIGIBILITY:
Inclusion Criteria:

1. 281 obese adolescents who participated in the randomized controlled interventional trial with low GI index diet
2. Willingness to give written consent

Exclusion Criteria:

1. Subjects who are allergic to any ingredients listed in G-NiiB®, microbiome immunity formula.
2. Subjects with any condition that the investigator deems as a sound reason (e.g. active gastrointestinal diseases and malignancies) for disqualification from enrollment into the study.

Ages: 25 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
proportion of subjects achieving 5% weight loss | 24 weeks
  Proportion of subjects achieving 5% weight loss is a standard measurement for weight management using probiotics/prebiotics.
changes in BMI | 24 weeks
changes in body weight | 24 weeks
changes in waist circumference | 24 weeks

IPD SHARING:
Plan to Share IPD: No